CLINICAL TRIAL: NCT03417232
Title: Biologically Guided Flap Stability: the Role of Periosteum Retention on the Performance of the Coronally Advanced Flap. A Double Blind Randomized Clinical Trial
Brief Title: Biologically Guided Flap Stability: the Role of Periosteum Retention on the Performance of the Coronally Advanced Flap
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Siena (Other)
Responsible Party: Principal Investigator, Prof. Marco Ferrari, Full Professor, University of Siena
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAF0001
Record Dates: First submitted 2018-01-23; First posted 2018-01-31 (Actual); Last update posted 2018-02-01 (Actual); Status verified 2018-01

CONDITIONS: Gingival Recession, Localized
Keywords: gingival recession; coronally advanced flap; complete root coverage; flap elevation; flap thickness
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Split Full Split Elevation of CAF (Experimental): The central portion of the flap apical to the recession was elevated full thickness by the use of a small periostium elevator inserted into the probable sulcus
  Interventions: Procedure: CAF
- Split Elevation of CAF (Sham Comparator): The flap was fully elevated with a split thickness approach: the blade of the knife was inserted into the sulcus
  Interventions: Procedure: CAF

INTERVENTIONS:
Procedure: CAF — The design of the flap consisted of two horizontal beveled incisions (3mm in length) and two slightly oblique beveled incisions. The resulting trapezoidal-shaped flap was elevated in the coronal-apical direction. The suture of the flap started with two interrupted periosteal sutures performed at the most apical extension of the vertical releasing incisions; afterwards, it proceeded coronally with other interrupted sutures, each of them directed, from the flap to the adjacent buccal soft tissue, in the apical-coronal direction. The last sling suture allowed for the stabilization of the surgical papillae over the inter-dental connective tissue bed and allowed for a precise adaptation of the flap margin over the underlying convexity of the crown.

SUMMARY:
Aim: to evaluate the possible benefit on wound healing and flap stability of periosteum inclusion, comparing a "split-full-split" thickness flap elevation versus a "split" thickness approach performed during CAF for the treatment of isolated-type gingival recessions in the upper jaw.

Material and Methods: forty patients were randomized, 20 were treated with "split-full-split" (test group) and 20 with a "split" approach (control group). Analyzed parameters at 1 year were: CRC, percentage of Recession Coverage (RC), Keratinized tissue (KT) gain, patient-related outcome measurements.

DETAILED DESCRIPTION:
Treatment of buccal gingival recession (GR) is the common clinical requirement from patients who are mainly concerned about aesthetics. Noteworthy are also requests linked to root sensitivity, difficulty in oral hygiene procedures, presence of root caries and non-carious cervical lesions. GR defects, when left untreated, do not improve spontaneously and may progress toward increased recession depth (RD) and clinical attachment loss which increase the patient's aesthetic concern and the clinical discomfort due to augmented dental hypersensitivity.

Complete root coverage (CRC) can be considered the primary clinical outcome and selecting the surgical technique depends mainly on the local anatomical characteristics and on the patient's demands.

In patients with a residual amount of keratinized tissue apical to the recession defect, the coronal advanced flap (CAF) may be recommended. This surgical technique results in optimal root coverage, good color blending of the treated area with respect to adjacent soft tissues and a complete recovery of the original (pre-surgical) soft tissue marginal morphology. Furthermore, post-operative morbidity is reduced to a single area of surgical intervention and the overall chair time is limited.

When utilizing CAF technique, critical factors in CRC have been described in the literature. Flap positioning coronal to the CEJ and a tension-free flap design are among the most important ones. Moreover, flap thickness has been shown to influence the clinical outcomes of CAF procedure .

Coronally advanced flap has been widely validated by the literature for the treatment of single recession defects and, currently, different flap designs and technical modifications are available to clinicians.

De Sanctis and Zucchelli have recently introduced the "split-full-split" flap elevation modality. According to the authors, the modulation of flap thickness, produced by the inclusion of periosteum in the central area, increases flap thickness in the portion of the flap residing over the previously exposed avascular root surface. This, in turn, would give better stability to the flap. However, the partial-thickness flap approach is still commonly performed in the clinical practice and it is validated in the literature.

To date, evidence is still lacking on the influence of including the periosteum in the flap when compared with a split thickness approach in obtaining a CRC.

Thus, the aim of this double blind, controlled and randomized clinical trial was to evaluate the possible benefit on wound healing and flap stability of periosteum inclusion comparing a "split-full-split" flap elevation versus a "split" thickness approach when CAF is performed for the treatment of isolated-type gingival recessions in the upper jaw.

ELIGIBILITY:
Inclusion Criteria:

* age >18 years,
* no systemic diseases or pregnancy,
* smoking ≤10 cigarettes/day,
* full-mouth plaque score and full-mouth bleeding score ≤20%,
* presence of at least one Miller class I or II isolated recession defect (Miller, 1985) in the upper jaw and at least 2 mm of keratinized tissue apical to the recession,
* recession depth (RD) equal to or greater than 2mm,
* identifiable cemento-enamel junction (CEJ),
* vital teeth, free from caries or prosthetic crown,

Exclusion Criteria:

* systemic diseases or pregnancy,
* history of periodontal surgery at experimental sites.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-04-01 (Actual); Primary Completion 2015-04-30 (Actual); Study Completion 2015-04-30 (Actual)

PRIMARY OUTCOMES:
CRC | 12 months
  Percentages of recession with a Complete Root Coverage

SECONDARY OUTCOMES:
RC | 12 months
  percentages of Recession Coverage
KTH | 12 months
  Keratinized Tissue Height in mm.
VAS discomfort | 12 months
  patient's discomfort expressed in a 10 cm Visual Analogue Scale, indicating discomfort from 0 (no discomfort) to 10 (maximum discomfort)
VAS esthetic | 12 months
  patient's esthetic expressed in a 10 cm Visual Analogue Scale, indicating esthetic from 0 (worst esthetic) to 10 (optimum esthetic).
VAS satisfaction | 12 months
  patient's satisfaction expressed in a 10 cm. Visual Analogue Scale, indicating satisfaction from 0 (no satisfaction) to 10 (good satisfaction).

CONTACTS AND LOCATIONS:
Overall Officials: Massimo De Sanctis, MD, Principal Investigator — University of Siena

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Clementini M, Discepoli N, Danesi C, de Sanctis M. Biologically guided flap stability: the role of flap thickness including periosteum retention on the performance of the coronally advanced flap-A double-blind randomized clinical trial. J Clin Periodontol. 2018 Oct;45(10):1238-1246. doi: 10.1111/jcpe.12998. Epub 2018 Sep 14. PMID 30099762